CLINICAL TRIAL: NCT00575588
Title: A 52-Week International, Multi-centre, Randomized, Parallel-group, Double-blind, Active-controlled, Phase III Study With a 52-Week Extension Period to Evaluate the Safety and Efficacy of Saxagliptin in Combination With Metformin Compared With Sulphonylurea in Combination With Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Metformin Therapy Alone.
Brief Title: 52-week add-on to Metformin Comparison of Saxagliptin and Sulphonylurea, With a 52-week Extension Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1680C00001; EudraCT number 2007-003998-55
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2010-09-06 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 Inhibitors; HbA1c; incretins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sulfonylurea Compounds; saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin (Experimental)
  Interventions: Drug: Metformin; Drug: Saxagliptin
- Glipizide (Experimental)
  Interventions: Drug: Metformin; Drug: Sulphonylurea

INTERVENTIONS:
Drug: Metformin — open-label metformin
Drug: Sulphonylurea — Glipizide 5-20 mg capsules (titrated to optimal effect or highest tolerable dose during 18 weeks)
  Arms: Glipizide
Drug: Saxagliptin — Saxagliptin 5 mg tablets
  Other Names: Onglyza
  Arms: Saxagliptin

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to assess the efficacy and tolerability of saxagliptin in addition to metformin and compare to sulphonylurea in addition with metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes,
* Treatment with metformin alone on stable doses of 1500 mg or higher per day for at least 8 weeks prior to Visit 1,
* HbA1c >6.5% and ≤10.0%

Exclusion Criteria:

* Type 1 diabetes,
* history of diabetic ketoacidosis or hyperosmolar non-ketonic coma,
* Insulin therapy within one year of enrolment (with the exception of insulin therapy during a hospitalization or use in gestational diabetes)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 891 (Actual)
Dates: Start 2007-12; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Goke, Principal Investigator — University of Munich, Germany; Peter Ohman, MD, Study Director — AstraZeneca; Deborah Price, MSc, Study Chair — AstraZeneca
Locations (94):
- Finland (7):
  - Research Site, Hanko
  - Research Site, Helsinki
  - Research Site, Kuopio
  - Research Site, Kuusankoski
  - Research Site, Mikkeli
  - Research Site, Oulu
  - Research Site, Tampere
- Germany (17):
  - Research Site, Aschaffenburg
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, Mannheim
  - Research Site, Mülheim
  - Research Site, Pirna
  - Research Site, Ratzeburg
  - Research Site, Reinfeld
  - Research Site, Rhaunen
  - Research Site, Schmiedeberg
  - Research Site, Tübingen
  - Research Site, Wahlstedt
  - Research Site, Weinheim
- Hungary (12):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Gyula
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Székesfehérvár
- India (4):
  - Research Site, Bangalore, Karnataka
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Mumbai, Mashatra
  - Research Site, Jaipur, Rajasthan
- Netherlands (11):
  - Research Site, 's-Hertogenbosch
  - Research Site, Beek en Donk
  - Research Site, Deurne
  - Research Site, Dordrecht
  - Research Site, Losser
  - Research Site, Nijverdal
  - Research Site, Rijswijk
  - Research Site, Roelofarendsveen
  - Research Site, Rotterdam
  - Research Site, The Hague
  - Research Site, Volendam
- Norway (12):
  - Research Site, Bergen
  - Research Site, Elverum
  - Research Site, Flatåsen
  - Research Site, Hamar
  - Research Site, Hønefoss
  - Research Site, Inderoy
  - Research Site, Oslo
  - Research Site, Rådal
  - Research Site, Skedsmokorset
  - Research Site, Sogndal
  - Research Site, Spikkestad
  - Research Site, Trollåsen
- Russia (5):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Slovakia (6):
  - Research Site, Dolný Kubín
  - Research Site, Kosice - Tahanovce
  - Research Site, Moldava nad Bodvou
  - Research Site, Ružomberok
  - Research Site, Trnava
  - Research Site, Žilina
- South Korea (6):
  - Research Site, Wŏnju, Gangwon-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
- United Kingdom (13):
  - Research Site, Annan, Dumfries and Galloway
  - Research Site, Whitstable, Kent
  - Research Site, Hamilton, Lanarkshire
  - Research Site, Salford, Manchester
  - Research Site, Crawley, West Sussex
  - Research Site, Bradford-on-Avon, Wiltshire
  - Research Site, Blackpool
  - Research Site, Coatbridge
  - Research Site, Coventry
  - Research Site, Glasgow
  - Research Site, Motherwell
  - Research Site, Newcastle
  - Research Site, Sheffield
- Research Site, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Cook W, Minervini G, Bryzinski B, Hirshberg B. Saxagliptin efficacy and safety in patients with type 2 diabetes mellitus stratified by cardiovascular disease history and cardiovascular risk factors: analysis of 3 clinical trials. Postgrad Med. 2014 Oct;126(6):19-32. doi: 10.3810/pgm.2014.10.2818. PMID 25414932
- [Derived] Mintz ML, Minervini G. Saxagliptin versus glipizide as add-on therapy to metformin: assessment of hypoglycemia. Curr Med Res Opin. 2014 May;30(5):761-70. doi: 10.1185/03007995.2014.880674. Epub 2014 Jan 30. PMID 24397584
- [Derived] Goke B, Gallwitz B, Eriksson JG, Hellqvist A, Gause-Nilsson I. Saxagliptin vs. glipizide as add-on therapy in patients with type 2 diabetes mellitus inadequately controlled on metformin alone: long-term (52-week) extension of a 52-week randomised controlled trial. Int J Clin Pract. 2013 Apr;67(4):307-16. doi: 10.1111/ijcp.12119. PMID 23638466

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 891 participants were enrolled in the study; 33 participants did not enter the treatment period; 858 participants were randomized and treated.
Groups:
- Saxagliptin + Metformin: Saxagliptin 5 mg tablets added on to open-label metformin
- Glipizide + Metformin: Glipizide 5-20 mg capsules (titrated to optimal effect or highest tolerable dose during 18 weeks) added on to open-label metformin
Period: Overall Study
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Started | 428 (Randomized and treated) | 430 (Randomized and treated)
Completed | 165 (Completed 104 weeks of treatment) | 147 (Completed 104 weeks of treatment)
Not Completed | 263 | 283
Not completed — Adverse Event | 11 | 13
Not completed — Withdrawal by Subject | 27 | 31
Not completed — Lost to Follow-up | 1 | 3
Not completed — Death | 4 | 2
Not completed — Incorrect enrollment | 8 | 4
Not completed — Study specific discontinuation criteria | 203 | 218
Not completed — Severe non-compliance to protocol | 5 | 7
Not completed — Safety reasons | 2 | 1
Not completed — Elevated triglyceride | 1 | 0
Not completed — Patient moved | 1 | 3
Not completed — Impossible to determine HbA1c | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin | Total
Number analyzed (Participants) | 428 | 430 | 858
Age Continuous [Mean (Standard Deviation); unit: years] | 57.50 (10.26) | 57.59 (10.37) | 57.55 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 216 | 198 | 414
  Male | 212 | 232 | 444

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (HbA1c) Change From Baseline to Week 52
Description: Adjusted mean change from baseline in HbA1c achieved with saxagliptin added on to metformin versus glipizide added on to metformin at Week 52 (Per Protocol Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated as the Week 52 value minus the baseline value.
Time Frame: Baseline to 52 Weeks
Population: Randomized participants who completed the 52 weeks of treatment had both baseline and week 52 HbA1c measurement and had no significant protocol deviations
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 293 | 293
Percent
  Baseline | 7.46 (0.045) | 7.53 (0.045)
  Week 52 | 6.74 (0.042) | 6.71 (0.042)
  Adjusted Change from Baseline to Week 52 | -0.74 (0.038) | -0.80 (0.038)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.05 to 0.16], Standard Error of Mean 0.053

2. Secondary Outcome: Proportion of Participants Reporting at Least One Episode of Any Hypoglycaemic Event Over 52 Weeks
Description: Proportion of participants reporting at least one episode of any hypoglycaemic event for saxagliptin added on to metformin versus glipizide added on to metformin over 52 weeks (Safety Analysis Set)
Time Frame: From Baseline to Week 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 428 | 430
Percentage of Participants | 3 [-38.1 to -28.5] | 36.3 [0 to 0]
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; p < 0.0001, Fisher Exact — Between group comparison significant after controlling overall alpha of the study; Mean Difference (Net) = -33.2, 95% CI 2-sided [-38.1 to -28.5]

3. Secondary Outcome: Body Weight Change From Baseline to Week 52
Description: Adjusted mean change from baseline in Body Weight achieved with saxagliptin added on to metformin versus glipizide added on to metformin at Week 52 (Safety Analysis Set). Body Weight is a continuous measure, the change from baseline for each participant is calculated as the Week 52 (LOCF) value minus the baseline value.
Time Frame: Baseline, Week 52 (Last Observation Carried Forward)
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in the LOCF analysis, participants must have had a baseline and at least 1 post-baseline measurement
Measure: Mean (Standard Error); unit: kilogram
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 424 | 426
kilogram
  Baseline | 88.7 (0.91) | 88.6 (0.95)
  Week 52 | 87.6 (0.90) | 89.7 (0.99)
  Adjusted Change from Baseline to Week 52 | -1.1 (0.17) | 1.1 (0.17)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Between group comparison significant after controlling overall alpha of the study; Mean Difference (Net) = -2.2, 95% CI [-2.7 to -1.7], Standard Error of Mean 0.24

4. Secondary Outcome: Mean Slope of the Regressions of Change From Week 24 to Week 52 in HbA1c
Description: Mean slopes of regression of change from Week 24 to Week 52 in HbA1c for saxagliptin added on to metformin versus glipizide added on to metformin (Per Protocol Analysis Set) achieved by fitting a mixed model with subject specific slopes for the time effect (weeks on randomized treatment was utilized). This analysis gives an assessment of the durability of the HbA1c effect.
Time Frame: Week 24 to Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 289 | 293
Percent | 0.001 (0.001) | 0.004 (0.001)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — Between group comparison significant after controlling overall alpha of the study; Mean Difference (Net) = -0.002, 95% CI 2-sided [-0.0046 to -0.0001], Standard Error of Mean 0.001

5. Other Pre Specified Outcome: Hemoglobin A1c (HbA1c) Change From Baseline to Week 104
Description: Adjusted mean change from baseline in HbA1c achieved with saxagliptin added on to metformin versus glipizide added on to metformin at Week 104 (Full Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated as the Week 104 value minus the baseline value.
Time Frame: Baseline, Week 104
Population: Number of subjects with observed values at Week 104 was n=184 for saxagliptin + metformin and n=160 for glipizide + metformin
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 423 | 423
Percent
  Baseline | 7.65 (0.044) | 7.65 (0.041)
  Week 104 | 7.27 (0.050) | 7.27 (0.046)
  Adjusted Change from Baseline to Week 104 | -0.41 (0.041) | -0.35 (0.043)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; Repeated Measures; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.17 to 0.06], Standard Error of Mean 0.059

6. Other Pre Specified Outcome: Proportion of Participants Reporting at Least One Episode of Any Hypoglycaemic Event Over 104 Weeks
Description: Proportion of participants reporting at least one episode of any hypoglycaemic event for saxagliptin added on to metformin versus glipizide added on to metformin over 104 weeks (Safety Analysis Set)
Time Frame: Baseline, Week 104
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 428 | 430
Percentage of Participants | 3.5 | 38.4
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; Mean Difference (Net) = -34.9, 95% CI 2-sided [-39.8 to -30.0]

7. Other Pre Specified Outcome: Body Weight Change From Baseline to Week 104
Description: Adjusted mean change from baseline in Body Weight achieved with saxagliptin added on to metformin versus glipizide added on to metformin at Week 104. Body Weight is a continuous measure, the change from baseline for each participant is calculated as the Week 104 value minus the baseline value.
Time Frame: Baseline, Week 104
Population: Number of subjects with observed values at Week 104 was n=186 for saxagliptin + metformin and n=165 for glipizide + metformin
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 424 | 426
kilograms
  Baseline | 88.69 (0.905) | 88.57 (0.955)
  Week 104 | 87.47 (0.898) | 89.80 (0.987)
  Adjusted Change from Baseline to Week 104 | -1.47 (0.200) | 1.29 (0.205)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; Repeated Measures; Mean Difference (Net) = -2.76, 95% CI 2-sided [-3.32 to -2.20], Standard Error of Mean 0.286

8. Other Pre Specified Outcome: Mean Slope of the Regressions of Change From Week 24 to Week 104 in HbA1c
Description: Mean slopes of regression of change from Week 24 to Week 104 in HbA1c for saxagliptin added on to metformin versus glipizide added on to metformin (Full Analysis Set) achieved by fitting a mixed model with subject specific slopes for the time effect (weeks on randomized treatment was utilized). This analysis gives an assessment of the durability of the HbA1c effect.
Time Frame: Week 24 to Week 104
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Number analyzed (Participants) | 373 | 377
Percent | 0.0041 (0.0005) | 0.0076 (0.0005)
Statistical Analysis 1: Comparison: Saxagliptin + Metformin vs Glipizide + Metformin; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Net) = -0.0035, 95% CI 2-sided [-0.0048 to -0.0022], Standard Error of Mean 0.0007

ADVERSE EVENTS:
Arm/Group | Saxagliptin + Metformin | Glipizide + Metformin
Serious Adverse Events (participants affected / at risk) | 54/428 | 55/430
Other Adverse Events (participants affected / at risk) | 105/428 | 201/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Saxagliptin + Metformin (N=428) | Glipizide + Metformin (N=430)
Atrial Fibrillation (Cardiac disorders) | 2 | 2
Coronary Artery Disease (Cardiac disorders) | 2 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Atrioventricular Block Complete (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 1
Myocardial Ischemia (Cardiac disorders) | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Fibrillation (Cardiac disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 2
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Coronary Artery Occlusion (Cardiac disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Anal Abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Helicobacter Gastritis (Infections and infestations) | 0 | 1
Superinfection (Infections and infestations) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Lesion (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 1
Open Wound (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastasis To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Salivary Gland Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Acute Abdomen (Gastrointestinal disorders) | 0 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Allergy To Arthropod Sting (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal Edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Deafness Bilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Biliary Colic (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Cerebrovascular Disorder (Nervous system disorders) | 1 | 0
Cerebral Ischemia (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Ischemic Stroke (Nervous system disorders) | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Aortic Aneurysm (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Herpes Zoster Ophthalmic (Infections and infestations) | 1 | 0
Salmonella Sepsis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Biliary Tract Infection (Infections and infestations) | 0 | 1/420
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bronchial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lip Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumor Ulceration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Transient Ischemic Attack (Nervous system disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Rectal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 0
Retinal Vein Occlusion (Eye disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 1
Device Malfunction (General disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 3
Hyperthyroidism (Endocrine disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Circulatory Collapse (Vascular disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin + Metformin (N=428) | Glipizide + Metformin (N=430)
Diarrhoea (Gastrointestinal disorders) | 25 | 17
Nasopharyngitis (Infections and infestations) | 46 | 41
Hypoglycaemia (Metabolism and nutrition disorders) | 15 | 165
Upper Respiratory Tract Infection (Infections and infestations) | 25 | 16
Hypertension (Vascular disorders) | 19 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No